CLINICAL TRIAL: NCT07266558
Title: A Phase 4, Randomized, Observer-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of mRNA-1283 And mRNA-1273 Variant-Containing Formulation in Adults 50 to 64 Years of Age Without Underlying Conditions That Put Them at High Risk for Severe Outcomes From COVID-19
Brief Title: A Study to Evaluate the Efficacy and Safety of mRNA-1283 and mRNA-1273 in Participants 50 to 64 Years of Age Without High-Risk Conditions for Severe Coronavirus Disease 2019 (COVID-19)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: mRNA-1273_1283-P401
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1283; SARS-CoV-2; mRNA vaccine; Coronavirus; Messenger RNA; COVID-19; COVID-19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- mRNA-1273 (Variant Formulation) (Experimental): Participants will receive a single intramuscular (IM) injection of mRNA-1273 on Day 1.
  Interventions: Biological: mRNA-1273
- mRNA-1283 (Variant Formulation) (Experimental): Participants will receive a single IM injection of mRNA-1283 on Day 1.
  Interventions: Biological: mRNA-1283
- Placebo (Placebo Comparator): Participants will receive a single IM injection of placebo on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: mRNA-1273 (Variant Formulation)
Biological: mRNA-1283 — Sterile liquid for injection
  Arms: mRNA-1283 (Variant Formulation)
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mRNA-1283 and mRNA-1273 (variant formulations) in adults 50 to 64 years of age without high risk factors for severe COVID-19.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy and without underlying medical conditions that may put them at higher risk of experiencing severe outcomes of COVID-19, as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.

Key Exclusion Criteria:

* History of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection within 3 months prior to enrollment.
* Acutely ill or febrile within 72 hours prior to or at the Screening Visit or Day 1.
* Receipt of any of the following:

  * COVID-19 vaccine within 3 months prior to enrollment,
  * Any licensed non COVID-19 vaccine within 28 days before or planned receipt within 28 days after the study intervention, except an influenza vaccine, which may be given 14 days before or after receipt of the study intervention,
  * Corticosteroids at ≥10 milligrams (mg)/day of prednisone or equivalent for >14 days in total within 90 days prior to Day 1 or is anticipating the need for corticosteroids at any time during the study or,
  * Systemic immunosuppressive treatment within 180 days prior to the Screening or is anticipating the need for systemic immunosuppressive treatment at any time during participation in the study.
* Has donated ≥450 mL of blood products within 28 days prior to the Screening Visit or plans to donate blood products within 28 days post study injection.
* Has participated in an investigational clinical study within 28 days prior to the Screening Visit based on the medical history interview or plans to do so while participating in this study.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30000 (Estimated)
Dates: Start 2025-11-26 (Actual); Primary Completion 2027-06-16 (Estimated); Study Completion 2027-06-16 (Estimated)

PRIMARY OUTCOMES:
VE of mRNA-1273 (Variant Formulation) to Prevent the First Event of Symptomatic COVID-19 after Study Injection | Day 1 through Day 181
  The VE is defined as the percent reduction in the hazard of the first event of symptomatic COVID-19 after study injection (each vaccine arm versus placebo) and will be estimated using 1-hazard ratio (HR).
Vaccine Efficacy (VE) of mRNA-1283 (Variant Formulation) to Prevent the First Event of Symptomatic COVID-19 after Study Injection | Day 1 through Day 181
  The VE is defined as the percent reduction in the hazard of the first event of symptomatic COVID-19 after study injection (each vaccine arm versus placebo) and will be estimated using 1-hazard ratio (HR).
Number of Participants with Unsolicited Adverse Events (AEs) | Day 1 through Day 28
Number of Participants with Serious AEs (SAEs), Medically Attended AEs (MAAEs), AEs of Special Interest (AESIs), and AEs Leading to Discontinuation | Day 1 through Day 181

SECONDARY OUTCOMES:
Number of Participants with a First Event of Severe COVID-19 after Study Injection | Day 1 through Day 181

CONTACTS AND LOCATIONS:
Locations (149):
- United States (149):
  - Accel Clinical Research, Birmingham, Alabama
  - Cullman Clinical Trials, Cullman, Alabama
  - AMR Clinical Mobile, Mobile, Alabama
  - Velocity Clinical Research, Mobile, Mobile, Alabama
  - Lenzmeier Family Medicine - Avacare, Glendale, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Velocity Clinical Research - Phoenix, Phoenix, Arizona
  - Foothills Research Center/Avacare, Phoenix, Arizona
  - Headlands Research Scottsdale, Scottsdale, Arizona
  - Fiel Family and Sports Medicine / Avacare, Tempe, Arizona
  - Avacare, Colton, California
  - CenExel CNR, Garden Grove, California
  - Velocity Clinical Research, Huntington Park, Huntington Park, California
  - Velocity Clinical Research - San Diego - ERN - PPDS-Site Number:8400010, La Mesa, California
  - Velocity Clinical Research - Los Angeles, Los Angeles, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Velocity Clinical Research -- Banning, San Bernardino, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Tekton Research, LLC, Denver, Colorado
  - Tekton Research, LLC, Fort Collins, Colorado
  - Critical Care, Pulmonary and Sleep Associates, P.LLP/Avacare, Lakewood, Colorado
  - Tekton Research, LLC, Longmont, Colorado
  - New England Research Associates, Bridgeport, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Velocity Clinical Research-Washington, DC, Washington D.C., District of Columbia
  - Hillcrest Medical Research, LLC, DeLand, Florida
  - University Clinical Research-Deland, LLC d/b/a Accel Research Sites - Deland Clinical Research Unit, DeLand, Florida
  - Suncoast Research Associates, LLC, Doral, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - CenExel Research Centers of America, Hollywood, Florida
  - NextPhase Research Florida, Hollywood, Florida
  - Health Awareness Inc., Jupiter, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites - Lakeland Clinical Research Unit, Lakeland, Florida
  - Sandhill Research, LLC d/b/a Accel Research Sites- St. Pete-Largo Clinical Research Unit, Largo, Florida
  - Accel Research Sites, Maitland, Florida
  - Global Health Research Center, Inc., Miami Lakes, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Innovation Medical Research Center, Palmetto Bay, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Global Health Research Center, Inc., Tampa, Florida
  - Javara Inc. and PRIVIA Medical Group of Georgia, LLC, Albany, Georgia
  - DelRicht Research, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Accel Research Sites - Neurostudies, Decatur, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - Javara Inc. and Privia Medical Group of Georgia, LLC, Fayetteville, Georgia
  - Velocity Clinical Research Savannah, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Velocity Clinical Research - Boise - ERN - PPDS, Meridian, Idaho
  - DM Clinical Research - Melrose Park, Melrose Park, Illinois
  - Velocity Clinical Research Valparaiso, Valparaiso, Indiana
  - Velocity Clinical Research - Sioux City, Sioux City, Iowa
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Tekton Research, LLC, Wichita, Kansas
  - DelRicht Research, Louisville, Kentucky
  - Versailles Family Medicine - CCT Research, Versailles, Kentucky
  - Velocity Clinical Research-Baton Rouge, Baton Rouge, Louisiana
  - Velocity Clinical Research - Covington, Covington, Louisiana
  - Avacare, Kenner, Louisiana
  - Velocity Clinical Research, Lafayette, Lafayette, Louisiana
  - DelRicht Research, Mandeville, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Velocity Clinical Research, New Orleans, New Orleans, Louisiana
  - DelRicht Research, Prairieville, Louisiana
  - Annapolis Internal Medicine, Annapolis, Maryland
  - Centennial Medical Group, Columbia, Maryland
  - Velocity Clinical Research, Rockville, Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - DM Clinical Research - Brookline, Brookline, Massachusetts
  - ActivMed Practices & Research, LLC, Methuen, Massachusetts
  - Headlands Research Detroit, Southfield, Michigan
  - DM Clinical Research - Southfield, Southfield, Michigan
  - Javara Inc. and Mankato Clinic, Ltd., Mankato, Minnesota
  - Velocity Clinical Research Gulfport, Gulfport, Mississippi
  - Clinical Research Professionals, Chesterfield, Missouri
  - AMR Clinical, Kansas City, Missouri
  - Clay-Platte Family Medicine Clinic, Kansas City, Missouri
  - DelRicht Research, Springfield, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - DelRicht Research, Town and Country, Missouri
  - Avacare Research/Methodist Physicians Clinic, Fremont, Nebraska
  - Velocity Clinical Research, Grand Island, Grand Island, Nebraska
  - Velocity Clinical Research, Lincoln, Nebraska
  - Velocity Clinical Research Norfolk, Norfolk, Nebraska
  - Velocity Clinical Research Omaha, Omaha, Nebraska
  - Avacare/Midwest Regional Health Services, Omaha, Nebraska
  - Papillion Research/Avacare, Papillion, Nebraska
  - Santa Rosa Medical Centers of Nevada, Las Vegas, Nevada
  - DM Clinical Research - Jersey City, Jersey City, New Jersey
  - DM Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Velocity Clinical Research - Albuquerque, Albuquerque, New Mexico
  - Rochester Clinical Research, Rochester, New York
  - Velocity Clinical Research, Durham, Durham, North Carolina
  - Eximia Research - NC, LLC, Raleigh, North Carolina
  - TMA Headlands LLC d/b/a Trial Management Associates, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Velocity Clinical Research - Cleveland, Beachwood, Ohio
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research-Mt. Auburn, Cincinnati, Ohio
  - Velocity Clinical Research Springdale, Cincinnati, Ohio
  - Tekton Research, LLC, Edmond, Oklahoma
  - Tekton Research, LLC, Moore, Oklahoma
  - DelRicht Research, Tulsa, Oklahoma
  - Tekton Research, LLC, Yukon, Oklahoma
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Summit Headlands LLC, Portland, Oregon
  - Hatboro Medical Associates/Avacare, Horsham, Pennsylvania
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Velocity Clinical Research - East Greenwich, East Greenwich, Rhode Island
  - Velocity Clinical Research, Anderson, Anderson, South Carolina
  - DelRicht Research, Charleston, South Carolina
  - Velocity Clinical Research - Columbia, Columbia, South Carolina
  - Coastal Carolina Research Center, LLC, North Charleston, South Carolina
  - Velocity Clinical Research Spartanburg, Spartanburg, South Carolina
  - Velocity Clinical Research Union, Union, South Carolina
  - DelRicht Research, Hendersonville, Tennessee
  - Velocity Clinical Research, Abilene, Abilene, Texas
  - Tekton Research, LLC, Austin, Texas
  - Velocity Clinical Research - Austin, Austin, Texas
  - Tekton Research, LLC, Beaumont, Texas
  - Javara Inc. and Privia Medical Group Gulf Coast, PLLC, Conroe, Texas
  - Velocity Clinical Research - Dallas, Dallas, Texas
  - Avacare, Fort Worth, Texas
  - DM Clinical Research - Houston, Houston, Texas
  - DelRicht Research, Prosper, Texas
  - Be Well Clinical Studies, Round Rock, Texas
  - DM Clinical Research - San Antonio, San Antonio, Texas
  - Tekton Research, LLC, San Antonio, Texas
  - Javara Inc. and Privia Medical Group Gulf Coast, PLLC, San Marcos, Texas
  - Javara Inc. and Privia Medical Group - North Texas, Stephenville, Texas
  - DM Clinical Research - Sugar Land, Sugar Land, Texas
  - Javara Inc. and Privia Medical Group Gulf Coast, PLLC, Sugar Land, Texas
  - Olympus Clinical Research, Sugar Land, Texas
  - DM Clinical Research - Tomball, Tomball, Texas
  - Cope Family Medicine / Avacare, Bountiful, Utah
  - Mountain View/Avacare, Pleasant View, Utah
  - JBR Clinical Research, Salt Lake City, Utah
  - Olympus Family Medicine/Avacare, Salt Lake City, Utah
  - J. Lewis Research, Inc/Jordan River Family Medicine, South Jordan, Utah
  - South Ogden Family Medicine/ Avacare, South Ogden, Utah
  - Velocity Clinical Research - Salt Lake City (West Jordan), West Jordan, Utah
  - Charlottesville Medical Research, LLC, Charlottesville, Virginia
  - Velocity Clinical Research-Hampton, Hampton, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - Velocity Clinical Research - Suffolk, Suffolk, Virginia
  - Velocity Clinical Research, Spokane, Spokane, Washington